CLINICAL TRIAL: NCT00978328
Title: A Prospective, Multi-center, Observational Registry of Patients Using Prescription Medications Containing Oxycodone Immediate Release for the Treatment of Pain
Brief Title: Oxycodone User Registry (OUR)
Status: Completed | Type: Observational
Sponsor: Ortho-McNeil Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Vice President, Medical Affairs, Internal Medicine
Other Study IDs: CR015670
Record Dates: First submitted 2009-09-15; First posted 2009-09-16 (Estimated); Last update posted 2010-04-02 (Estimated); Status verified 2010-04

CONDITIONS: Pain
Keywords: Pain conditions; Oxycodone immediate release; Percocet®, Tylox®; Roxicodone®; Registry; Side effects; Observational; Pain management
MeSH Terms: conditions — Pain; Agnosia | interventions — Oxycodone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- 001: oxycodone immediate release (OXYRX) Characteristics of pts. receiving prescription medications containing OXYRX
  Interventions: Drug: oxycodone immediate release (OXYRX)

INTERVENTIONS:
Drug: oxycodone immediate release (OXYRX) — Characteristics of pts. receiving prescription medications containing OXYRX

SUMMARY:
The purpose of this study is to describe clinical and demographic characteristics of patients receiving prescription medications containing oxycodone immediate release (OXYRX), to characterize patient and prescriber perceptions of the effectiveness outcomes and tolerability of OXYRX treatment, to describe prescriber decision-making about pain management with a Schedule II opioid and to explore how prescribers identify suspected abuse of pain medications.

DETAILED DESCRIPTION:
Real-world utility of Schedule II immediate release opioids depends on both efficacy and side effects. Few existing data sources systematically captured opioid-related side effects and their impact on patient outcomes and physician practice. This study is expected to lead to an in-depth understanding of patient and prescriber perceptions of both effectiveness and side effects associated with medications containing the most widely prescribed oral Schedule II immediate release opioid for pain management, oxycodone immediate release (OXYRX), alone (eg, Roxicodone®) or in combination (eg, Percocet®, Tylox®) in actual clinical practice. This is a prospective, multi-center, observational patient registry. Adult outpatients who have pain due to a non-cancerous condition meeting study eligibility will be enrolled. Prescribers will treat patients according to their usual practice. Prescribers will treat patients, meeting study eligibility, with OXYRX according to their usual practice.

ELIGIBILITY:
Inclusion Criteria:

* Pain requiring treatment with a Schedule II immediate release opioid within 3 days following the baseline visit
* and pain that warrants treatment with a prescription for OXYRX PRN (alone or in combination) for at least 5 days after the baseline visit

Exclusion Criteria:

* Use of any Schedule II opioid within 30 days prior to informed consent
* planned use of other opioids (Schedule II-V) while using OXYRX
* malignancy other than superficial skin cancers (ie, basal cell, squamous cell) within the past year

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting for treatment of a painful condition with a Schedule II opioid at an outpatient setting will be potential candidates for enrollment for this registry.
Sampling Method: Non-Probability Sample
Enrollment: 827 (Actual)
Dates: Start 2009-06; Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Describe clinical / demographic characteristics of patients receiving OXYRX; characterize patient / prescriber perceptions of the effectiveness outcomes and tolerability of OXYRX treatment; describe prescriber decision-making about pain meds | Baseline, Day 1, Day 3, Day 7, Day 14, Day 21, Day 28

CONTACTS AND LOCATIONS:
Overall Officials: Ortho-McNeil Janssen Scientific Affairs, LLC Clinical Trial, Study Director — Ortho-McNeil Janssen Scientific Affairs, LLC